CLINICAL TRIAL: NCT04790591
Title: Is Partial Knee Replacement as Same-day Surgery Generalizable? A Non-selective Interventional Study on Efficacy, Patient Satisfaction, and Safety in a Public Hospital Setting
Brief Title: Is Partial Knee Replacement as Same-day Surgery Generalizable?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Magnus Tveit, Orthopaedic consultant, PhD, Region Skane
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02000
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Same-day Surgery
Keywords: Arthroplasty, PKR, Same-day discharge, Same-day surgery, UKA
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Intervention Model Description: Open clinical trial with a subgroup analysis
  (One can argue whether this study should be defined as a cohort study or as an open clinical trial. The idea of the study originated from the need to observe/confirm the feasibility and safety aspects of a routine which as of today has become common practice, namely same-day surgery, but as such it may also be categorized as a treatment... Either way, based on the preselection of age and comorbidity often reported in the literature, a two-arm subgroup analysis of the nonselective study participants will be conducted.)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Age <80 yrs. and ASA class <3 (Active Comparator): To follow a same-day surgery protocol when undergoing a partial knee replacement procedure.
  Interventions: Procedure: Same-day surgery
- Age ≥80 yrs. and/or ASA class ≥3 (Active Comparator): To follow a same-day surgery protocol when undergoing a partial knee replacement procedure.
  Interventions: Procedure: Same-day surgery

INTERVENTIONS:
Procedure: Same-day surgery — To be allowed same-day discharge certain postoperative criteria have to be met. These are categorized into four dimensions - vital parameters, urinary function, bleeding, and mobilization.

SUMMARY:
Fast-track/rapid recovery/Enhanced Recovery After Surgery (ERAS) programs have proven both safe and effective in joint replacement surgery, to the degree where same-day surgery have been tested in selected cases. A transition of the minor partial knee replacement (PKR) procedure, compared with the alternative and more commonly used total knee replacement (TKR) for knee osteoarthritis, into a same-day regime seems reasonable. Especially as PKR is reported to have lower risk of short-term complications than does TKR.

The aim of this study is to assess efficacy, patient satisfaction and safety outcome measures for PKR when using a same-day surgery protocol in a Swedish healthcare context where ERAS programs nowadays are considered common ground.

With no preselection of patients, all PKR cases by one high-volume surgeon will chronologically be scheduled as the first morning case for one consecutive year, and thereby be included in the study. In order for discharge, strict post-surgery criteria will have to be met.

The thesis is that the same-day surgery will be both feasible and safe.

DETAILED DESCRIPTION:
The eligibility for being considered a medial PKR is either antero-medial osteoarthritis or spontaneous osteonecrosis of the knee. The study-protocol has a pragmatic approach to whom of the PKR candidates will be considered for same-day surgery, as no preselection of patients will be done prior to surgery. I.e., everyone considered for a PKR procedure will be informed prior to surgery by a multidisciplinary team (anesthesiologist, nurse, physiotherapist, and surgeon) that if the surgery will be scheduled in the morning, he/she will then be following a same-day surgery protocol and likely be discharged to home later the same day.

All of one high-volume surgeon´s (MT) first morning slots for one consecutive year will be dedicated to patients who will undergo PKR surgery, and thereby also be included in the study. The slots will be filled continuously as the patients are put up for surgery. When all slots have been taken within one week any additional PKR cases will be assigned to surgery later in the day the same week (as will all the THRs and the TKRs during this period) and consequently not taking part in this study. The operation scheduling will be put together on a weekly basis, in a strict chronological order, by a team of nurses without any insight from the surgeon in question.

The criteria for discharge will be based strictly on postoperative parameters categorized into four dimensions - vital parameters, urinary function, bleeding, and mobilization. The vital parameters will be measured and scored by the National Early Warning Score (NEWS), where the threshold for discharge will be conservatively set to zero (NEWS 0). The urinary function algorithm for discharge will, in short, be if no need for catheterization and less than 200 ml of residual volume after spontaneous void. A compression stocking will be removed six hours post-surgery and if no ongoing bleeding discharge can be considered. Last, but not least, a physiotherapist will evaluate whether basic activity of daily living (ADL) can be performed in a safely manner using crutches.

Primary outcome measures for this three-month follow-up will be safety, i.e. number of adverse events and readmissions. Secondary aims will be feasibility such as same-day surgery achievement and extra outpatient visits needed and for what reasons. Patient-satisfaction will also be evaluated after the participants/patients have ben discharged to their own home. A two-arm subgroup analysis will be conducted between those aged <80 yrs and classified as ASA <3 and those aged ≥80 yrs. and/or classified as ASA class ≥3.

Descriptive data will be presented as unadjusted means with standard deviations (SD), medians with range, or as numbers with proportions (%). The between-group differences will be presented as means with 95% confidence intervals (95% CI) and p values using Welch's test, Mann-Whitney U-test and Likelihood Ratio Test (or when violated Fisher's exact test) for numerical, ordinal and categorical variables respectively. Multivariate analyses will be conducted using logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* All participants/patients that will undergo a partial knee replacement (PKR) procedure within one consecutive year by one high-volume surgeon (i.e. no preselection of patients will be made)

Exclusion Criteria:

* PKR procedures performed by other surgeons
* One-stage bilateral PKR procedures
* PKR procedures not given the first surgery slot of the day

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Safety - adverse events and/or readmissions | 3 months
  Number of severe complications that may have had a causal association with the same-day surgery and any readmissions, no matter the cause

SECONDARY OUTCOMES:
Feasibility - same-day surgery discharge and resources relocated from the inpatient to the outpatient department | 12 hours and 3 months respectively
  Number of participants that will achieve discharge on the day of surgery and number of additional outpatient visits required compared to planned
Patient-satisfaction | 24 hours
  Number of participants that will agree on all three of the following statements when phoned the day after surgery: "A positive experience; would do it again; can recommend to others"

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Tveit, MD, PhD, Principal Investigator — Region Skane
Locations (2):
- Sweden (2):
  - Skåne University Hospital, Lund, Region Skåne
  - Trelleborg Hospital, Trelleborg, Region Skåne

IPD SHARING:
Plan to Share IPD: No